CLINICAL TRIAL: NCT01339091
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Dalbavancin to a Comparator Regiment (Vancomycin and Linezolid) for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Efficacy and Safety of Dalbavancin for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUR001-301
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Abscess; Wound Infection; Surgical Site Infection; Cellulitis
MeSH Terms: conditions — Abscess; Wound Infection; Surgical Wound Infection; Cellulitis | interventions — dalbavancin; Vancomycin; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dalbavancin (Experimental)
  Interventions: Drug: Dalbavancin
- Vancomycin with possible switch to oral linezolid (Active Comparator)
  Interventions: Drug: Vancomycin / Linezolid

INTERVENTIONS:
Drug: Dalbavancin — IV Dalbavancin 1000 mg on Day 1 and 500 mg on Day 8
  Arms: Dalbavancin
Drug: Vancomycin / Linezolid — IV Vancomycin (1 gram Q 12 hours or 15mg/Kg Q 12 hours) with optional switch to oral linezolid (600 mg Q12 hours). Total duration of therapy is 10-14 days.
  Arms: Vancomycin with possible switch to oral linezolid

SUMMARY:
The primary object is to compare the early clinical efficacy (after 48-72 hours of therapy) of dalbavancin to the comparator regimen (vancomycin with the option to switch to oral linezolid) for the treatment of patients with a suspected or proven gram-positive bacterial skin or skin structure infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 - 85 years of age.
2. Signed and dated informed consent document.
3. Major abscess, surgical site infection, traumatic wound infection or cellulitis suspected or confirmed to be caused by Gram-positive bacteria.
4. At least two (2) local signs and symptoms of ABSSSI and at least one (1) systemic sign of infection.
5. Requires a minimum of 3 days of IV therapy.
6. Patient willing and able to comply with study procedures.

Exclusion Criteria:

Patients presenting with any of the following:

1. A contra-indication to any required study drug.
2. Pregnant or nursing females.
3. Sustained shock.
4. Participation in another study of an investigational drug or device within 30 days.
5. Receipt of a systemically or topically administered antibiotic within 14 days prior to randomization, except receipt of a single dose of a short-acting antibacterial drug 3 or more days prior to randomization.
6. Infection due to a dalbavancin or vancomycin-resistant organism.
7. Evidence of meningitis, necrotizing fasciitis, gas gangrene, gangrene, septic arthritis, osteomyelitis, and/or endovascular infection.
8. Exclusively gram-negative bacterial or a fungal ABSSSI.
9. Venous catheter infection.
10. Infection of a diabetic foot ulcer or a decubitus ulcer.
11. Device-related infections.
12. Gram-negative bacteremia.
13. Infected burns.
14. Infected limb with critical ischemia.
15. Superficial/simple skin and skin structure infections.
16. Concomitant condition requiring non-study antibacterial therapy.
17. ABSSSI requiring therapy for longer than 14 days.
18. Adjunctive therapy with hyperbaric oxygen.
19. More than 2 surgical interventions for ABSSSI anticipated.
20. Chronic inflammatory condition precluding assessment of clinical response.
21. Absolute neutrophil count < 500 cells/mm3.
22. Human immunodeficiency virus (HIV) infection with a CD4 cell count < 200 cells/mm3.
23. Recent bone marrow transplant, > 20 mg prednisolone per day (or equivalent) or receiving immunosuppressant drugs after organ transplantation.
24. Regular, chronic antipyretic use in patients unable to modify during the first three days of study drug therapy.
25. Life expectancy less than 3 months.
26. Conditions that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.
27. Prior participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunne, MD, Study Director — Durata Therapeutics Inc., an affiliate of Allergan plc
Locations (83):
- United States (53):
  - Durata Study Site, Anaheim, California
  - Durata Study Site, Azusa, California
  - Durata Study Site, Bellflower, California
  - Durata Study Site, Buena Park, California
  - Durata Study Site, Carmel, California
  - Durata Study Site, Chula Vista, California
  - Durata Study Site, Covina, California
  - Durata Study Site, Fountain Valley, California
  - Durata Study Site, La Mesa, California
  - Durata Study Site, Long Beach, California
  - Durata Study Site, Los Alamitos, California
  - Durata Study Site, Los Angeles, California
  - Durata Study Site, Oceanside, California
  - Durata Study Site, Palm Desert, California
  - Durata Study Site, Pasadena, California
  - Durata Study Site, Sacramento, California
  - Durata Study Site, San Diego, California
  - Durata Study Site, Santa Ana, California
  - Durata Study Site, Sylmar, California
  - Durata Study Site, Torrance, California
  - Durata Study Site, Upland, California
  - Durata Study Site, Whittier, California
  - Durata Study Site, Miami, Florida
  - Durata Study Site, Orlando, Florida
  - Durata Study Site, Saint Cloud, Florida
  - Durata Study Site, Tampa, Florida
  - Durata Study Site, Columbus, Georgia
  - Durata Study Site, Savannah, Georgia
  - Durata Study Site, Idaho Falls, Idaho
  - Durata Study Site, Pocatello, Idaho
  - Durata Study Site, Moline, Illinois
  - Durata Study Site, Rock Island, Illinois
  - Durata Study Site, Baton Rouge, Louisiana
  - Durata Study Site, Lafayette, Louisiana
  - Durata Clinical Site, New Orleans, Louisiana
  - Durata Study Site, Opelousas, Louisiana
  - Durata Study Site, Detroit, Michigan
  - Durata Study Site, Minneapolis, Minnesota
  - Durata Study Site, Las Vegas, Nevada
  - Durata Study Site, Somers Point, New Jersey
  - Durata Study Site, Buffalo, New York
  - Durata Study Site, Lake Success, New York
  - Durata Study Site, New Hyde Park, New York
  - Durata Study Site, Staten Island, New York
  - Durata Study Site, The Bronx, New York
  - Durata Study Site, Winston-Salem, North Carolina
  - Durata Study Site, Columbus, Ohio
  - Durata Study Site, Lima, Ohio
  - Durata Study Site, Toledo, Ohio
  - Durata Study Site, Pittsburgh, Pennsylvania
  - Durata Study Site, Houston, Texas
  - Durata Study Site, Madison, Wisconsin
  - Durata Study Site, Middleton, Wisconsin
- Canada (2):
  - Durata Study Site, Winnipeg, Manitoba
  - Durata Study Site, Trois-Rivières, Quebec
- Croatia (3):
  - Durata Study Site, Dubrovnik
  - Durata Clinical Site, Slavonski Brod
  - Durata Study Site, Zagreb
- Durata Clinical Site, Tbilisi, Georgia
- Germany (2):
  - Durata Study Site, Bochum
  - Durata Study Site, Münster
- Poland (4):
  - Durata Study Site, Krakow
  - Durata Study Site, Legionowo
  - Durata Study Site, Warsaw
  - Durata Study Site, Wroclaw
- Russia (11):
  - Durata Study Site, Kharkiv, Ukraine
  - Durata Study Site, Kyiv City, Ukraine
  - Durata Study Site, Moscow
  - Durata Clinical Site, Moscow
  - Durata Study Site, Perm
  - Durata Study Site, Saint Petersburg
  - Durata Clinical Site, Saint Petersburg
  - Durata Study Site, Saratov
  - Durata Study Site, Smolensk
  - Durata Study Site, Tomsk
  - Durata Study Site, Yekaterinburg
- Ukraine (7):
  - Durata Study Site, Cherkasy
  - Durata Study Site, Ivano-Frankivsk
  - Durata Study Site, Kharkiv
  - Durata Study Site, Kyiv
  - Durata Study Site, Uzhhorod
  - Durata Study Site, Zaporizhzhya
  - Durata Study Site, Zhytomyr

REFERENCES:
- [Derived] Gonzalez PL, Rappo U, Akinapelli K, McGregor JS, Puttagunta S, Dunne MW. Outcomes in Patients with Staphylococcus aureus Bacteremia Treated with Dalbavancin in Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):423-434. doi: 10.1007/s40121-021-00568-7. Epub 2021 Dec 14. PMID 34905144
- [Derived] Boucher HW, Wilcox M, Talbot GH, Puttagunta S, Das AF, Dunne MW. Once-weekly dalbavancin versus daily conventional therapy for skin infection. N Engl J Med. 2014 Jun 5;370(23):2169-79. doi: 10.1056/NEJMoa1310480. PMID 24897082

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalbavancin: Dalbavancin : IV Dalbavancin 1000 mg on Day 1 and 500 mg on Day 8
- Vancomycin +/- Oral Linezolid: Vancomycin : IV Vancomycin (dosed per standard of care) with optional switch to oral linezolid (600 mg Q12 hours). Total duration of therapy is 10-14 days.
Period: Overall Study
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Started | 288 | 285
Safety Population | 284 | 284
Completed | 261 | 257
Not Completed | 27 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid | Total
Number analyzed (Participants) | 288 | 285 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.3) | 48.9 (15.08) | 48.9 (15.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 112 | 230
  Male | 170 | 173 | 343

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Efficacy
Description: Clinical response at 48-72 hours post study drug initiation, based on measurements of acute bacterial skin and skin structure infections (ABSSSI) lesion size and temperature
Time Frame: 48-72 hours after the initiation of study therapy
Population: The ITT population consisted of all randomly assigned patients regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Number analyzed (Participants) | 288 | 285
participants
  Clinical Responder | 240 | 233
  Clinical Non-Responder | 48 | 52
Statistical Analysis 1: Comparison: Dalbavancin vs Vancomycin +/- Oral Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test is a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the 95% CI for the difference in response rates in the ITT population is greater than -10% the NI of dalbavancin to vancomycin/linezolid will be concluded; Difference in Proportions = 1.5, 95% CI 2-sided [-4.6 to 7.9] — Confidence intervals were adjusted for fever at baseline

2. Secondary Outcome: >= 20% Reduction in Lesion Area
Description: Clinical response at 48-72 hours post study drug initiation, based on measurements of acute bacterial skin and skin structure infections (ABSSSI) lesion size
Time Frame: 48-72 hours after the initiation of study therapy
Population: The ITT population consisted of all randomly assigned patients regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Number analyzed (Participants) | 288 | 285
participants
  Clinical Responder | 259 | 259
  Clinical Non-Responder | 29 | 26

3. Secondary Outcome: Clinical Status
Description: Compare the clinical efficacy at end of treatment visit of dalbavancin to the comparator regimen based on lesion size, local signs, temperature and receipt of non-study antibiotics
Time Frame: End of Treatment Visit (Day 14-15)
Population: Clinical Evaluable Population based on certain inclusion/exclusion criteria, length of study therapy, concomitant antibacterials, concomitant surgical procedure and non-missing data.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Number analyzed (Participants) | 246 | 243
participants
  Clinical Success | 214 | 222
  Clinical Failure | 32 | 21

4. Secondary Outcome: Clinical Status
Description: Compare the clinical efficacy at the day 28 follow-up visit of dalbavancin to the comparator regimen based on lesion size, local signs, temperature and receipt of non-study antibiotics
Time Frame: Follow-Up Visit (day 28)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Number analyzed (Participants) | 226 | 229
participants
  Clinical Success | 212 | 220
  Clinical Failure | 14 | 9

ADVERSE EVENTS:
Time Frame: Begins from the time that the patient provides informed consent through the last follow up visit, Day 70. Any SAE occurring any time after the reporting period must be promptly reported if a causal relationship to investigational product is suspected.
Description: Adverse events were analyzed in the safety population which is defined as all patients in the ITT population who received at least 1 dose of dalbavancin or vancomycin (active) study drug.
Arm/Group | Dalbavancin | Vancomycin +/- Oral Linezolid
Serious Adverse Events (participants affected / at risk) | 5/284 | 12/284
Other Adverse Events (participants affected / at risk) | 36/284 | 54/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalbavancin (N=284) | Vancomycin +/- Oral Linezolid (N=284)
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Embolic pneumonia (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalbavancin (N=284) | Vancomycin +/- Oral Linezolid (N=284)
Headache (Nervous system disorders) | 14 | 14
Nausea (Gastrointestinal disorders) | 12 | 13
Hypertension (Vascular disorders) | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 11
Vomiting (Gastrointestinal disorders) | 3 | 6
Asthenia (General disorders) | 1 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide Durata an opportunity to review any proposed publication or other type of disclosure at least 30 days before they are submitted. If any patent action is required to protect intellectual property rights, the Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days. If the study is part of a multi-center study, the Investigator agrees that the first publication is to be a joint publication covering all centers.